CLINICAL TRIAL: NCT05332184
Title: Cardiac T1 Mapping Enables Risk Prediction of LV Dysfunction After Surgery for Aortic Regurgitation
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Martin Sinn, Resident, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: BAV_T1
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Aortic Regurgitation
MeSH Terms: conditions — Aortic Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients prior to aortic valve surgery
  Interventions: Procedure: aortic valve surgery

INTERVENTIONS:
Procedure: aortic valve surgery

SUMMARY:
To assess whether cardiac T1 mapping for detection of myocardial fibrosis enables preoperative identification of patients at risk for early left ventricular dysfunction after surgery of aortic regurgitation.

DETAILED DESCRIPTION:
We hypothesized that a diffuse interstitial myocardial fibrosis may be present in AR patients who experience early systolic LV dysfunction after aortic valve surgery. We aimed to evaluate the association between preoperative cardiac T1 mapping for detection of myocardial fibrosis and early systolic LV dysfunction after surgery for aortic regurgitation.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with severe aortic regurgitation referred for aortic valve surgery were prospectively enrolled in the study.

Exclusion Criteria:

* history of coronary artery disease
* acute aortic valve disease (i.e., type A aortic dissection or infectious endocarditis)
* common contraindications for MRI such as severe obesity and metallic foreign bodies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 40 consecutive AR patients referred for aortic valve surgery were included.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Native T1 | baseline (Prior surgery)
  Measured with MRI

IPD SHARING:
Plan to Share IPD: Undecided
IPD can be shared anonymized upon reasonable request.